CLINICAL TRIAL: NCT05023616
Title: Evaluation of Efficacy of Online Real-time Home CPR Training Program : a Randomized Open-label Clinical Trial
Brief Title: Evaluation of Efficacy of Online Real-time Home CPR Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki Jeong Hong, Clinical associate professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-2107-205-1239
Record Dates: First submitted 2021-08-06; First posted 2021-08-26 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Cardiopulmonary Resuscitation; Cardiopulmonary Arrest; Education
Keywords: Cardiopulmonary Resuscitation; Education
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time home CPR training (Experimental): Online real-time home CPR(cardiopulmonary resuscitation) training will be provided to participants
  Interventions: Other: Real-time home CPR training
- Conventional CPR training (Active Comparator): Conventional CPR training will be provided to participants
  Interventions: Other: Conventional CPR training

INTERVENTIONS:
Other: Real-time home CPR training — The participants in the intervention group will have Little Anne QCPR mannequins (Laerdal, Stavanger, Norway) delivered to their homes. The participants will use an online platform specifically developed for CPR training (HEROS Remote app). The training program will provide video-based self-instruction training followed by hands-on chest compression training with the instructor. The hands-on chest compression training session provides real-time chest compression quality measurement followed by real-time feedback from the instructor. Chest compression quality will be measured by Little Anne QCPR mannequins.
  Arms: Real-time home CPR training
Other: Conventional CPR training — Participants in the conventional CPR training program group will be provided CPR education with the "Home Education and Resuscitation Outcome Study (HEROS)" program that is currently provided in Seoul, Korea. The HEROS program is a 1-hour training course, consisting of a 30-minute video-based self-instruction training with a mannequin. The program also includes a bystander CPR simulation with a simulated dispatcher using the participants own cell phone. Little Anne QCPR mannequins will be provided to measure and give feedback on the participants chest compression performance.
  Arms: Conventional CPR training

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a real-time home CPR(cardiopulmonary resuscitation) training program. The study participants will be allocated to two different CPR training programs. The intervention group will participate in the real-time home CPR training program while the control group will participate in the conventional CPR training program. The investigators will compare the quality of chest compression between the two study groups. The investigators hypothesize that the new real-time home CPR training program is non-inferior to the preexisting conventional CPR training program.

DETAILED DESCRIPTION:
Bystander CPR(cardiopulmonary resuscitation) is important for the survival of out-of-hospital cardiac arrest patients. CPR training for the general public is important to improve the rate and quality of bystander CPR. Conventional CPR education was conducted under face-to-face contact with instructors and multiple trainees gathered at a training center, but after the coronavirus disease 2019 pandemic, face-to-face training became difficult. To overcome this limitation the investigators have developed a new real-time home CPR training program. The training program delivers Little Anne QCPR mannequins (Laerdal, Stavanger, Norway) to each participants homes and the participants use an application specifically developed for CPR training that automatically connects wirelessly to the Little Anne QCPR mannequin through Bluetooth so that the instructor can give real-time feedback on chest compression quality to participants.

The purpose of this study is to evaluate the effectiveness of a real-time home CPR(cardiopulmonary resuscitation) training program. The study participants will be allocated to two different CPR training programs. The intervention group will participate in the real-time home CPR training program while the control group will participate in the conventional CPR training program. The investigators will compare the quality of chest compression between the two study groups. Chest compression quality at the start of both training programs and after completion of the programs will be measured by Little Anne QCPR mannequins used in the training programs. The investigators hypothesize that the new real-time home CPR training program is non-inferior to the preexisting conventional CPR training program.

ELIGIBILITY:
Inclusion Criteria:

* Adults without prior CPR training within 6 months

Exclusion Criteria:

* Healthcare providers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Average compression depth | Immediately after the training program has been completed, participants will be asked to perform chest compression for 2 minutes. The outcome measure will be collected from the 2 minutes of chest compression at this point.
  Average compression depth of chest compression performed for 2 minutes

SECONDARY OUTCOMES:
Proportion of adequate compression depth | Immediately after the training program has been completed, participants will be asked to perform chest compression for 2 minutes. The outcome measure will be collected from the 2 minutes of chest compression at this point.
  Proportion of adequate compression depth performed for 2 minutes
Average compression rate | Immediately after the training program has been completed, participants will be asked to perform chest compression for 2 minutes. The outcome measure will be collected from the 2 minutes of chest compression at this point.
  Average compression rate of chest compression performed for 2 minutes
Proportion of adequate compression rate | Immediately after the training program has been completed, participants will be asked to perform chest compression for 2 minutes. The outcome measure will be collected from the 2 minutes of chest compression at this point.
  Proportion of adequate compression rate performed for 2 minutes
No-flow fraction | Immediately after the training program has been completed, participants will be asked to perform chest compression for 2 minutes. The outcome measure will be collected from the 2 minutes of chest compression at this point.
  Proportion of no-flow time during 2 minutes of chest compression

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jeong Hong, MD, Study Chair — Department of Emergency Medicine, Seoul National University Hospital; STEPHEN GW LEE, MD, Principal Investigator — Department of Emergency Medicine, SMG-SNU Boramae Medical Center; Seulki Choi, MD, Principal Investigator — Department of Emergency Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Background] Nolan JP, Monsieurs KG, Bossaert L, Bottiger BW, Greif R, Lott C, Madar J, Olasveengen TM, Roehr CC, Semeraro F, Soar J, Van de Voorde P, Zideman DA, Perkins GD; European Resuscitation Council COVID-Guideline Writing Groups. European Resuscitation Council COVID-19 guidelines executive summary. Resuscitation. 2020 Aug;153:45-55. doi: 10.1016/j.resuscitation.2020.06.001. Epub 2020 Jun 7. PMID 32525022
- [Background] Cheng A, Magid DJ, Auerbach M, Bhanji F, Bigham BL, Blewer AL, Dainty KN, Diederich E, Lin Y, Leary M, Mahgoub M, Mancini ME, Navarro K, Donoghue A. Part 6: Resuscitation Education Science: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S551-S579. doi: 10.1161/CIR.0000000000000903. Epub 2020 Oct 21. No abstract available. PMID 33081527
- [Background] Nas J, Thannhauser J, Vart P, van Geuns RJ, Muijsers HEC, Mol JQ, Aarts GWA, Konijnenberg LSF, Gommans DHF, Ahoud-Schoenmakers SGAM, Vos JL, van Royen N, Bonnes JL, Brouwer MA. Effect of Face-to-Face vs Virtual Reality Training on Cardiopulmonary Resuscitation Quality: A Randomized Clinical Trial. JAMA Cardiol. 2020 Mar 1;5(3):328-335. doi: 10.1001/jamacardio.2019.4992. PMID 31734702
- [Background] Park GJ, Kong SYJ, Song KJ, Shin SD, Kim TH, Ro YS, Myklebust H, Birkenes TS. The Effectiveness of a New Dispatcher-Assisted Basic Life Support Training Program on Quality in Cardiopulmonary Resuscitation Performance During Training and Willingness to Perform Bystander Cardiopulmonary Resuscitation: A Cluster Randomized Controlled Study. Simul Healthc. 2020 Oct;15(5):318-325. doi: 10.1097/SIH.0000000000000435. PMID 32604135